CLINICAL TRIAL: NCT02737657
Title: Observational, Prospective, Parallel Cohort Study to Evaluate Tolerability of Canagliflozin and Sulphonylurea on a Background Therapy of Metformin With or Without a DPP-4 Inhibitor During Ramadan Fasting in Patients With Type 2 Diabetes
Brief Title: An Observational Study to Evaluate Tolerability of Canagliflozin and Sulphonylurea in Type 2 Diabetes Patients During Ramadan
Acronym: CRATOS
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108100; 28431754DIA4016 (Other: Janssen-Cilag International)
Record Dates: First submitted 2016-03-23; First posted 2016-04-14 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Canagliflozin; Metformin; Diabetes Mellitus, Type 2; INVOKANA; Sulfonylurea
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cohort 1: Participants who are already receiving Canagliflozin and Metformin with or without a DPP-4 inhibitor daily during Ramadan period will be observed as the part of study.
- Cohort 2: Participants who are already receiving any sulphonylurea and Metformin with or without a DPP-4 inhibitor daily during Ramadan period will be observed as a part of study.

SUMMARY:
The primary purpose of this study is to describe the tolerability of canagliflozin and any sulphonylurea (each administered with metformin with or without a DPP-4 inhibitor), in terms of the percentage of patients with at least one episode of hypoglycaemia, in patients with T2DM who fast during Ramadan.

DETAILED DESCRIPTION:
This is non-randomized, parallel-cohort, prospective, multicenter (when more than one hospital works on a medical research study), observational study to describe the treatment of T2DM with canagliflozin during the Holy Month of Ramadan. Observed participants will be participants with T2DM (at the time of enrollment) who are being treated with either canagliflozin or any sulphonylurea, each administered on a background therapy of metformin with or without a DPP-4 inhibitor within clinical practice, and who intend to fast during the Ramadan period. On enrollment, patients will enter one of two parallel treatment cohorts based on their ongoing T2DM therapy: canagliflozin and metformin with or without a DPP-4 inhibitor will be the treatment of interest, while any sulphonylurea and metformin with or without a DPP-4 inhibitor will serve as the reference standard treatment. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who has a confirmed diagnosis of type 2 diabetes for more than 12 months before enrollment
* Participants who has been treated with canagliflozin or any sulphonylurea, each on a background therapy of metformin with or without a dipeptidyl peptidase 4 (DPP-4) inhibitor, for >12 weeks before enrollment
* Participants Intends to fast during Ramadan in 2016
* Participants Will be able to continue on the products under study (i.e., canagliflozin or any sulphonylurea, each with metformin with or without a DPP-4 inhibitor) through the Ramadan period, as judged by the participating physician
* Participants who has a glycated hemoglobin (HbA1c) measurement less than and equal to (<=) 8.5% within 8 weeks before the start of Ramadan.

Exclusion Criteria:

* Participant is being treated with insulin and/or any type 2 diabetes mellitus (T2DM) therapy other than canagliflozin, any sulphonylurea, and metformin with or without a DPP 4 inhibitor, or has changed their T2DM therapy within 12 weeks before enrollment (dose changes of canagliflozin, a sulphonylurea, metformin, and a DPP 4 inhibitor where applicable are accepted)
* Participant is currently being treated with loop diuretics
* Participants who has a history of severe hypoglycaemia events within the 6 months prior to enrollment (defined as a hypoglycaemia event for which the patient required assistance from another person, or which resulted in seizure or loss of consciousness).
* Participants who has heart failure (NYHA 3-4) or advanced cardiovascular disease.
* Participants who has an estimated glomerular filtration rate (eGFR) less than (<) 60 milliliter/minute (mL/min)/1.73 m^2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a confirmed diagnosis of type 2 diabetes and has been treated with canagliflozin or any sulphonylurea, each on a background therapy of metformin with or without a DPP-4 inhibitor, will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With at Least one Episode of Hypoglycaemia | during the Ramadan period (up to 1 month)
  Hypoglycaemia events are defined by symptoms (e.g., dizziness, visual blurring, palpitations, nausea, sweating, confusion, tremor or intense hunger) reported by the patient in the patient diary, with confirmation by a physician where applicable; Episode may be documented via a self-monitored blood glucose measurement <70 milligram/deciliter (mg/dl).

SECONDARY OUTCOMES:
Number of Participants With Volume Depletion Events | during the Ramadan period (up to 1 month)
Treatment Adherence Based on the Percentage of Prescribed Doses of Canagliflozin or Sulphonylurea Taken by Participants | during the Ramadan period (up to 1 month)
Time to the First Hypoglycaemia Event | during the Ramadan period (up to 1 month)
Relationship of Hypoglycaemia Events With Clinical Parameters | during the Ramadan period (up to 1 month)
  Precipitating factors, symptoms and blood glucose concentration during hypoglycaemia episode will be described.
Relationship of Hypoglycaemia Events With Used Treatment | during the Ramadan period (up to 1 month)
  Causal relationship of hypoglycaemia event to treatment will be evaluated.
Relationship of Hypoglycaemia Events With Treatment Adherence | during the Ramadan period (up to 1 month)
  Treatment adherence will be based on the percentage of prescribed doses of canagliflozin or sulphonylurea that are missed during the Ramadan period, as reported in the patient diary. Any changes in study medication (i.e. missed or delayed dosing) due to hypoglycaemia events will be captured.
Relationship of Hypoglycaemia Events With Number of Fasting Days | during the Ramadan period (up to 1 month)
  Number of days when fasting was broken due to hypoglycaemia or hypoglycaemia prevention will be captured.
Relationship of Volume Depletion Events With Clinical Parameters | during the Ramadan period (up to 1 month)
  Precipitating factors, symptoms and blood glucose concentration during volume depletion related adverse events will be described.
Relationship of Volume Depletion Events With Used Treatment | during the Ramadan period (up to 1 month)
  Causal relationship of volume depletion related adverse event to treatment will be evaluated.
Relationship of Volume Depletion Events With Treatment Adherence | during the Ramadan period (up to 1 month)
  Treatment adherence will be based on the percentage of prescribed doses of canagliflozin or sulphonylurea that are missed during the Ramadan period, as reported in the patient diary. Any changes in study medication (i.e. missed or delayed dosing) due to Volume depletion related adverse events will be captured.
Relationship of Volume Depletion Events With Number of Fasting Days | during the Ramadan period (up to 1 month)
  Number of days when fasting was broken due to the volume depletion related adverse event will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (9):
- Kuwait City, Kuwait
- Lebanon (6):
  - Amioûn
  - Beirut
  - Nabatieh
  - Saida
  - Taalabya
  - Tripoli
- United Arab Emirates (2):
  - Al Ain City
  - Dubai

REFERENCES:
- [Derived] Hassanein M, Echtay A, Hassoun A, Alarouj M, Afandi B, Poladian R, Bennakhi A, Nazar M, Bergmans P, Keim S, Hamilton G, Azar ST. Tolerability of canagliflozin in patients with type 2 diabetes mellitus fasting during Ramadan: Results of the Canagliflozin in Ramadan Tolerance Observational Study (CRATOS). Int J Clin Pract. 2017 Oct;71(10):e12991. doi: 10.1111/ijcp.12991. Epub 2017 Aug 29. PMID 28851109